CLINICAL TRIAL: NCT00002659
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED STUDY TO EVALUATE THE EFFECT OF CISPLATIN/EPINEPHRINE INJECTABLE GEL (PRODUCT MPI 5010) WHEN ADMINISTERED INTRATUMORALLY FOR ACHIEVEMENT OF TREATMENT GOALS IN RECURRENT OR REFRACTORY SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK
Brief Title: Cisplatin Plus Epinephrine in Treating Patients With Recurrent or Refractory Head and Neck Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Matrix Pharmaceutical (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064225; MP-414-94-2; NCI-V95-0676
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

INTERVENTIONS:
Drug: cisplatin-e therapeutic implant

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if treatment with cisplatin plus epinephrine is effective for head and neck cancer.

PURPOSE: Randomized double-blinded phase III trial to determine the effectiveness of cisplatin plus epinephrine in injectable gel form in treating patients who have recurrent or refractory head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of intratumoral injection of a cisplatin/epinephrine gel (CDDP-e TI) to placebo gel for local control of recurrent or refractory squamous cell carcinoma of the head and neck. II. Assess achievement of a preselected (by the investigator) treatment goal for the most troublesome tumor in patients with recurrent or refractory squamous cell carcinoma of the head and neck following up to 6 weekly intratumoral treatments with CDDP-e TI vs. placebo gel. III. Compare the effect of CDDP-e TI to placebo gel on total local tumor volume per patient. IV. Evaluate the time to response and time to progression for the most troublesome tumor after local treatment with CDDP-e TI vs. placebo gel. V. Assess the improvement in or stabilization of quality of life in these patients as measured by the FACT-H&N questionnaire. VI. Compare the histopathology of injected lesions that respond to local treatment.

OUTLINE: Randomized, double-blind study. Randomization weighted 2:1 in favor of Arm I. Arm I: Intratumoral Chemotherapy. Cisplatin (NSC-119875) and Epinephrine in a bovine collagen gel, MP 5010, CDDP-e TI. Arm II: Control. NS in a bovine collagen gel, PLCB.

PROJECTED ACCRUAL: Up to 120 evaluable patients will be studied to provide 80 evaluable patients on Arm I and 40 evaluable patients on Arm II.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell carcinoma of the head and neck that is recurrent or refractory following at least 1 course of therapy Primary or metastatic tumors involving skin, nodes (palpable and biopsy- proven), subcutaneous tissue, or muscle allowed No involvement of major artery or any visceral organ Measurable lesions accessible for direct intratumoral injection with no immediate risk of hemorrhage or embolization Most troublesome tumor (identified by the investigator) at least 0.5 cc and no greater than 20 cc Smaller tumors eligible for treatment but not for efficacy assessment An improvable primary treatment goal (palliative or preventive) for most troublesome tumor must be identified by the investigator prior to enrollment If multiple tumors qualify as most troublesome and share the primary physician-selected treatment goal, the largest tumor is selected Patient may also select a most troublesome tumor and 1 palliative treatment goal for that tumor (need not match the physician-selected tumor or goal) No fibrotic lesions (e.g., previously irradiated lesion with no subsequent disease progression) No tumors involving or threatening to invade the carotid or other major vessel

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60%-100% Life expectancy: At least 6 months Hematopoietic: Absolute granulocyte count greater than 1,000/mm3 Platelet count greater than 75,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 1.5 times normal Cardiovascular: No NYHA class III/IV status No history of arrhythmia that would increase risk of treatment Other: No hypersensitivity to cisplatin, bovine collagen, epinephrine, or sulfites No significant history of extracranial carotid vascular disease from atherosclerosis, radiation therapy or previous carotid artery surgery No uncontrolled local infection at treatment sites No medical or psychiatric condition that would preclude informed consent No pregnant or nursing women Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: More than 28 days since any antineoplastic therapy or therapy with investigational agents Fully recovered from side effects of prior treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 1995-05

CONTACTS AND LOCATIONS:
Overall Officials: Mack H. Mabry, MD, Study Chair — SUGEN
Locations (28):
- United States (26):
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Comprehensive Cancer Center at JFK Medical Center, Atlantis, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Evanston Northwestern Health Care, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky College of Medicine, Lexington, Kentucky
  - Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - Creighton University Cancer Center, Omaha, Nebraska
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Boston Cancer Group, Memphis, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - University of Texas Southwestern Medical School, Dallas, Texas
  - Department of Otolaryngology, Milwaukee, Wisconsin
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Ville Marie Oncology Center, Montreal, Quebec